CLINICAL TRIAL: NCT00338767
Title: Depression Treatment to Improve Antiretroviral Adherence
Brief Title: Antidepressant Medication Plus Directly Observed Therapy for Improving Adherence to Antiretroviral Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Bangsberg, MD, Principal Investigator, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH063011 (NIH); R01MH063011 (NIH)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections; Depression
Keywords: AIDS; DOT; Directly Observed Therapy
MeSH Terms: conditions — HIV Infections; Depression; Acquired Immunodeficiency Syndrome; Directly Observed Therapy | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants receiving storefront directly observed therapy of anti-depressants (Fluoxetine)
  Interventions: Behavioral: Directly Observed Therapy (DOT); Drug: Fluoxetine
- Control (No Intervention): Participants receiving referral to mental health follow-up with the UCSF AIDS Health Project

INTERVENTIONS:
Behavioral: Directly Observed Therapy (DOT) — DOT includes storefront directly observed therapy of prescribed anti-depressants. Participants will meet with a study psychiatrist, who will prescribe an appropriate antidepressant medication. Subsequent meetings with the psychiatrist will occur weekly for the first 3 weeks, and then monthly for the duration of the study. Additionally, participants will have DOT visits every weekday morning for 1 month to take their antidepressant medications. After the first month, DOT visits will occur weekly or biweekly, depending on the medication regimen.
  Arms: Treatment
Drug: Fluoxetine — Medication treatment includes flouxetine for treatment of depression.
  Arms: Treatment

SUMMARY:
This study will evaluate the effectiveness of directly observed therapy plus antidepressant medication in improving adherence to antiretroviral drug therapy among HIV-infected homeless and marginally housed people with depression.

DETAILED DESCRIPTION:
Antiretroviral drug therapy (ART) is a type of medication treatment for HIV that impairs the virus's ability to multiply. When used properly, it has been shown to be successful in reducing HIV-related deaths. A 95% adherence rate to ART is required to adequately suppress the virus and prevent transmission. Low ART adherence rates are often linked to depression, which is especially common in HIV-infected homeless or marginally housed people. In these cases, treatment with antidepressant medication may be useful in improving ART adherence. Directly Observed Therapy (DOT), in which medication intake is closely monitored, is another method of enhancing treatment compliance. DOT improved treatment adherence during the tuberculosis epidemic of the 1990s, and is now gaining recognition as a model for improving ART adherence. This study will evaluate the effectiveness of combining DOT and antidepressant medication in improving ART adherence among HIV-infected homeless and marginally housed people with depression.

Participants in this 9-month, open-label study will be randomly assigned to a treatment group or a control group. The control group will be given the phone number of the University of California, San Francisco AIDS Health Project (AHP) to call and make an appointment with a psychiatrist. Participants who attend appointments will be evaluated to determine their mental health status. Participants who are deemed to benefit from treatment will be scheduled for regular appointments at the AHP, but will be responsible for administering their own medications. The treatment group will meet with a study psychiatrist, who will prescribe an appropriate antidepressant medication. Subsequent meetings with the psychiatrist will occur weekly for the first 3 weeks, and then monthly for the duration of the study. Additionally, participants will have DOT visits every weekday morning for 1 month to take their antidepressant medications. After the first month, DOT visits will occur weekly or biweekly, depending on the medication regimen. If an individual does not attend a visit, study staff will try to locate the individual in the neighborhood to deliver the medication. Medication for the weekend will be prepared by study staff, but participants will take it on their own at home. For the last 2 months of the study, DOT visits will occur once monthly, at which time participants will receive their entire month's supply of medication.

Participants in both groups will be asked to report to the study site weekly for 6 months and then monthly for the final 3 months to provide an update on the status of their housing, healthcare providers, case managers, and HIV medications. Additional interviews about housing, income, use of health services, drug use, sexual practices, and mental health will occur at the beginning of the study and three more times throughout the study. Blood tests will be performed monthly to assess viral load, and every 3 months to assess CD4 count. Participants taking HIV medications will be visited by study staff at home once a month so that use of HIV medications can be determined. At the end of the study, participants in the control group may continue receiving treatment at the AHP. Six months after the end of the study, participants in the treatment group may also begin treatment with a psychiatrist at the AHP.

ELIGIBILITY:
Inclusion Criteria:

* Homeless or marginally housed
* Score of greater than 13 on the Beck Depression Inventory (BDI)
* DSM-IV diagnosis of major depressive disorder, dysthymia, or minor depressive disorder
* Considered by the reviewing psychiatrist to benefit from antidepressant therapy
* Willing to take antidepressant medication or, if currently taking medication, willing to change medications if deemed appropriate
* Consents to coordinate with the primary medical provider
* Speaks English

Exclusion Criteria:

* Signs and symptoms consistent with diagnosis of dementia, as defined by DSM-IV
* Current substance abuse disorder requiring immediate residential or inpatient treatment
* At risk for suicide
* Presence of signs and symptoms consistent with psychotic depression, as defined by DSM-IV, warranting immediate hospitalization
* Any condition or use of any medication that may make simultaneous use of antidepressant medication unsafe
* Currently prescribed antidepressant therapy and in psychiatric treatment (treated by a psychiatrist within 3 months prior to study entry)
* Pregnant
* Bipolar disorder
* Current psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2001-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Improved depression scores | Measured at the end of 9 months

SECONDARY OUTCOMES:
HIV viral load | Measured monthly for 9 months
CD4 Count | Measured at baseline and Months 3, 6, and 9

CONTACTS AND LOCATIONS:
Overall Officials: David R. Bangsberg, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Market Street Study Site, San Francisco, California, United States

REFERENCES:
- [Derived] Grelotti DJ, Hammer GP, Dilley JW, Karasic DH, Sorensen JL, Bangsberg DR, Tsai AC. Does substance use compromise depression treatment in persons with HIV? Findings from a randomized controlled trial. AIDS Care. 2017 Mar;29(3):273-279. doi: 10.1080/09540121.2016.1226479. Epub 2016 Sep 2. PMID 27590273